CLINICAL TRIAL: NCT00367874
Title: Treatment of Polydrug-Using Opiate Dependents During Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSHF_ARA_001
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2006-08

CONDITIONS: Opiate Dependence; Drug Dependence; Substance Withdrawal Syndrome
Keywords: Opiate dependence; Benzodiazepine dependence; Polydrug Abuse; Detoxification; Withdrawal Treatment
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Substance Withdrawal Syndrome | interventions — Buprenorphine; Valproic Acid

INTERVENTIONS:
Drug: Buprenorphine
Drug: Valproate

SUMMARY:
Managed detoxification is a first and necessary step prior to treatment and rehabilitation. Detoxification can be a major obstacle for some patients, and the availability of managed and safe withdrawal is a prerequisite for long-term treatment.

In our clinical practice we have felt the need for a standardised and safe detoxification treatment regimen for our opioid addicts, as dependence on multiple drugs is so common.

Objectives

1. To assess whether a novel standardised treatment regimen - Buprenorphine (BPN) combined with Valproate (VPA) - will result in fewer withdrawal symptoms during detoxification of opiate-polydrug users than the existing treatment regimen, i.e. Clonidine (CLN) combined with Carbamazepine (CBZ).
2. To determine whether there are differences in treatment retention between the BPN/VPA and the CLN/CBZ groups.
3. To assess differences in clinical side-effects and biochemical interactions between the two treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

- Polydrug dependency (at least opiate and benzodiazepine dependency)

Exclusion Criteria:

* No severe psychiatric illness
* No history of epilepsy seizures
* No pregnancy or breastfeeding
* Fertile women must use contraceptives

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-02; Study Completion 2003-11

PRIMARY OUTCOMES:
Retention in treatment
Withdrawal symptoms

SECONDARY OUTCOMES:
Serum concentration of Valproate and Buprenorphine separately and in combination
Urine testing

CONTACTS AND LOCATIONS:
Overall Officials: Oistein Kristensen, MD, Principal Investigator — Sorlandet Hospital HF, Addiction Unit
Locations (1):
- Sorlandet Hospital HF, Addiction Unit (ARA), Kristiansand, Vest-Agder, Norway

REFERENCES:
- [Derived] Kristensen O, Lolandsmo T, Isaksen A, Vederhus JK, Clausen T. Treatment of polydrug-using opiate dependents during withdrawal: towards a standardisation of treatment. BMC Psychiatry. 2006 Nov 15;6:54. doi: 10.1186/1471-244X-6-54. PMID 17107609